CLINICAL TRIAL: NCT02967471
Title: Discovery of New Early Detection Biomarkers From Peripheral Blood of Acute Respiratory Distress Syndrome(ARDS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Principal Investigator, Hui Peng, Principal Investigator, The Third Affiliated Hospital of Southern Medical University
Other Study IDs: ARDS-ILC001
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ARDS group
- control group

SUMMARY:
Acute respiratory distress syndrome (ARDS) has a very poor prognosis and high mortality. To improve the early diagnosis of ARDS, there is an urgent need for novel biomarkers of ARDS. This project aims to detect novel biomarkers from peripheral blood , which can improve the early diagnosis and develop a more efficient therapy to enhance ARDS patient survival rate. Clinical data and blood sample were recorded before treatment and after treatment. Acute Physiology And Chronic Health Evaluation III (APACHE III) scores were calculated at enrolment. Different kinds of lymphocytes from blood samples would be detected by flow cytometry ,which could be used for discovering high sensitivity and specificity ARDS biomarker.

DETAILED DESCRIPTION:
Background Acute respiratory distress syndrome (ARDS) has a very poor prognosis and high mortality. To improve the early diagnosis of ARDS, there is an urgent need for novel biomarkers of ARDS. This project aims to detect novel biomarkers from peripheral blood , which can improve the early diagnosis and develop a more efficient therapy to enhance ARDS patient survival rate. Clinical data and blood sample were recorded before treatment and after treatment. Acute Physiology And Chronic Health Evaluation III (APACHE III) scores were calculated at enrolment. Different kinds of lymphocytes from blood samples would be detected by flow cytometry ,which could be used for discovering high sensitivity and specificity ARDS biomarker.

Eligibility Ages Eligible for Study: 18 years and older Genders Eligible for Study: Both Accepts Healthy Volunteers: Yes Sampling Method: Probility Samples

Study Population Patients who have ARDS and admitted in hospital

Primary Outcome Measures:

ILC2 and ILC3 number from peripheral blood of ARDS patients

Secondary Outcome Measures:

APACHE III score [ Time Frame: baseline, 1week, 2 weeks ] PaO2/FiO2 ratio[ Time Frame: baseline, 1week, 2 weeks ] Mortality or multi-organ failure [ Time Frame: 1 month ]

Groups:

1. Mild ARDS PaO2/FiO2=201～300 mmHg，and PEEP or CPAP≤5 cm
2. Moderate ARDS PaO2/FIO2=101～200 mmHg，and PEEP≥5 cm H2O
3. Severe ARDSPaO2/FIO2≤100 mmHg，and PEEP≥10 cm H2O
4. Healthy

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 years and older Genders Eligible for Study: Both Accepts Healthy Volunteers: Yes Sampling Method: Probility Samples Study Population：Patients who have ARDS and admitted in hospital Criteria：Inclusion Criteria:The Berlin definition of acute respiratory distress syndrome,ATS definition of severe pneumonia

Exclusion Criteria:

* age below 18 years,pregnancy,Expected survival under 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have ARDS and admitted in hospital
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
ILC 3 | 1 months after the onset
  innate lymphoid cells 3
ILC 2 | 1 months after the onset
  innate lymphoid cells 2

SECONDARY OUTCOMES:
APACHE III score | 1 months after the onset
PaO2/FiO2 ratio | 1 months after the onset
Mortality or multi-organ failure | 1 months after the onset

CONTACTS AND LOCATIONS:
Overall Officials: Jinhong Wang, M.D., Study Chair — The Third Affiliated Hospital of Southern Medical University; Hui Peng, M.M., Principal Investigator — The Third Affiliated Hospital of Southern Medical University; Hong Yang, M.D., Study Director — The Third Affiliated Hospital of Southern Medical University

IPD SHARING:
Plan to Share IPD: No